CLINICAL TRIAL: NCT06328777
Title: A Phase 1/2, Open-Label Study to Evaluate the Safety and Efficacy of Autologous CD19-specific Chimeric Antigen Receptor T Cells (CABA-201) in Subjects With Systemic Sclerosis
Brief Title: RESET-SSc: An Open-Label Study to Evaluate the Safety and Efficacy of CABA-201, a CD19-CAR T Cell Therapy, in Subjects With Systemic Sclerosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cabaletta Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAB-201-003
Record Dates: First submitted 2024-03-19; First posted 2024-03-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: CABA-201; autoimmune disease; anti-CD19 CAR-T therapy; systemic sclerosis; scleroderma
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Autoimmune Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CABA-201 (Experimental): Severe Skin Cohort: Infusion of CABA-201 with preconditioning in subjects with SSc with severe skin involvement
  Organ Cohort: Infusion of CABA-201 with preconditioning in subjects with SSc with organ involvement
  Interventions: Biological: CABA-201

INTERVENTIONS:
Biological: CABA-201 — Single intravenous infusion of CABA-201 at a single dose level following preconditioning with fludarabine and cyclophosphamide

SUMMARY:
RESET-SSc: A Phase 1/2 Open-Label Study to Evaluate the Safety and Efficacy of CABA-201, a CD19-CAR T cell therapy, in Subjects with Systemic Sclerosis

DETAILED DESCRIPTION:
Systemic sclerosis (SSc), also known as scleroderma , is a rare autoimmune disorder characterized by autoantibody production and abnormal B cell function. Though the cause of SSc is not well understood, it is thought to involve B cells that cause the body to attack different tissues in one's own body, causing skin and organ fibrosis. This study is being conducted to evaluate the safety and efficacy of an investigational therapy, CABA-201, a CD19-CAR T cell therapy, that can be given to patients with SSc who have active disease. A single dose of CABA-201 in combination with cyclophosphamide (CY) and fludarabine (FLU) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75
* A clinical diagnosis of SSc, based on the 2013 American College of Rheumatology and European League Against Rheumatism classification criteria.
* Early active disease
* Evidence of significant skin, pulmonary, renal, or cardiac involvement

Exclusion Criteria:

* Contraindication to leukapheresis
* History of anaphylactic or severe systemic reaction to fludarabine, cyclophosphamide or any of their metabolites
* Active infection requiring medical intervention at screening visit
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, psychiatric, cardiac, neurological, or cerebral disease, including severe and uncontrolled infections, such as sepsis and opportunistic infections.
* Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study, interfere with the assessment of the effects or safety of the investigational product or with the study procedures
* Severe lung or cardiac impairment
* Previous CAR T cell therapy
* Prior solid organ (heart, liver, kidney, lung) transplant or hematopoietic cell transplant

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate incidence of adverse events | Up to 28 days after CABA-201 infusion
  Incidence and severity of AEs

SECONDARY OUTCOMES:
To evaluate adverse events and laboratory abnormalities | Up to 156 weeks
  Incidence and severity of AEs, including changes in laboratory values and vital signs
To characterize the pharmacodynamics (PD) | Up to 156 weeks
  Levels of B cells in the blood
To characterize the pharmacokinetics (PK) | Up to 156 weeks
  Levels of CABA-201-positive T cells in the blood
To evaluate efficacy | Up to 156 weeks
  Proportion of subjects achieving revised CRISS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Cabaletta Bio
Locations (10):
- United States (10):
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No